CLINICAL TRIAL: NCT05548491
Title: A Two Stage, Multi-center, Vehicle-controlled, Study to Evaluate the Safety, Tolerability, and Pharmacodynamics of AZR-MD-001 and to Determine Common Symptoms in Contact Lens Discomfort (CLD)
Brief Title: Safety, Tolerability and Pharmacodynamics of AZR-MD-001 in Contact Lens Discomfort (CLD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Azura Ophthalmics (Industry)
Collaborators: Avania (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AZ202201
Record Dates: First submitted 2022-09-17; First posted 2022-09-21 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Contact Lens Discomfort

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: single-masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AZR-MD-001 1.0% (Experimental): AZR-MD-001 ointment/semi-solid drug (1.0%)
  Interventions: Drug: AZR-MD-001 ointment/semi-solid drug
- AZR-MD-001 vehicle (Placebo Comparator): AZR-MD-001 vehicle
  Interventions: Drug: AZR-MD-001 ointment/semi-solid drug

INTERVENTIONS:
Drug: AZR-MD-001 ointment/semi-solid drug — ointment/semi-solid drug

SUMMARY:
A two stage, multi-center, vehicle-controlled study to determine common symptoms in patients with Contact Lens Discomfort (CLD) in Stage 1 and to evaluate the safety, tolerability, and pharmacodynamics of AZR-MD-001 in Stage 2.

DETAILED DESCRIPTION:
A two stage, multi-center, vehicle-controlled study to determine common symptoms in patients with Contact Lens Discomfort (CLD) in Stage 1 and to evaluate the safety, tolerability, and pharmacodynamics of AZR-MD-001 in Stage 2.

For Stage 1 of the study, up to 12 participants who experience symptoms of CLD and experience concomitant meibomian gland dysfunction will complete a Screening visit followed by a hybrid concept elicitation and cognitive debriefing interview which can occur at the end of the Screening visit or up to 14 days later.

Stage 2 is a multi-center, single-masked, vehicle-controlled, randomized, parallel group study. Participants with CLD will be randomly assigned in a 1:1 ratio to receive either active AZR-MD-001 ointment/semi-solid drug (1.0%) or AZR-MD-001 vehicle for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of meibomian gland obstruction (based on a meibomian gland secretion (MGS) score of ≤12 for 15 glands of the lower lid) in both eyes.
* A history of wearing soft contact lenses for at least 6 months.
* Screening CLDEQ-8 score >12

Exclusion Criteria:

* Active ocular infection (bacterial, viral, or fungal).
* Participant is unlikely to follow study instructions or to complete all required study visit(s) or has a condition or situation that in the investigator's opinion, may put the participant at significant risk, may confound the study results, or may interfere significantly with the participant's participation in the study.
* Participant is an employee at the investigational site or is related to any member of the study staff.
* Participation in another clinical trial involving a therapeutic drug or device within the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2023-10-13 (Actual); Study Completion 2023-10-13 (Actual)

PRIMARY OUTCOMES:
Meibomian Glands Yielding Liquid Secretion (MGYLS) Yielding Liquid Secretion (MGYLS) | 3 months
  Change from baseline to month 3 in the number of Meibomian Glands Yielding Liquid Secretion (MGYLS)
Contact Lens Dry Eye Questionnaire-8 (CLDEQ-8) fluctuating vision | 3 months
  Change from baseline to month 3 in CLDEQ-8 fluctuating vision items. Scores can range from 0 (normal) to 9 (impacted vision).
  (summed responses to questions 3a and 3b only)
Contact Lens Dry Eye Questionnaire-8 (CLDEQ-8) total score | 3 months
  Change from baseline to month 3 in CLDEQ-8 total score. Scores can range from 0 (normal) to 37 (Impacted Contact Use).

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - University of New South Wales, School of Optometry and Vision Science, Sydney, New South Wales
  - Ophthalmic Trials Australia, Teneriffe, Queensland

IPD SHARING:
Plan to Share IPD: No